CLINICAL TRIAL: NCT00702806
Title: A Phase II, Open Label, Prospective, Randomized, Comparative Clinical Trial to Investigate the Appropriate Dose of a Single Injection of Org 36286 (Corifollitropin Alfa) to Initiate Multiple Follicular Growth in a Controlled Ovarian Hyperstimulation Protocol for IVF or IVF/ICSI.
Brief Title: Investigate Dose of Org 36286 to Initiate Multiple Follicular Growth in a Controlled Ovarian Hyperstimulation Protocol for IVF or IVF/ICSI (P07015)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07015; 38807
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Infertility; In Vitro Fertilization
Keywords: Pharmacological effects of drugs; Hormones; Hormone substitutes and Hormone Antagonists; Pharmacological Actions; Randomized; Multi-center; Multi-national
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; ganirelix; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Org 36286 120 μg + Puregon® 150 IU (Experimental): On Cycle Day 2 or Day 3, a single intra-abdominal injection of Org 36286 120 μg was administered to participants. On stimulation Day 8, a daily subcutaneous dose of Puregon® 150 IU was administered up to and including the time of Pregnyl® administration as a single dose of 10,000 IU subcutaneously. The maximum treatment duration of Puregon® 150 IU was 19 days. Orgalutran® 0.25 mg was administered subcutaneously once daily up to and including the day of Pregnyl®, when the leading follicle reached a size of >= 14 mm.
  Interventions: Drug: Org 36286; Drug: Puregon®; Drug: Orgalutran®; Drug: Pregnyl®
- Org 36286 180 μg + Puregon® 150 IU (Experimental): Cycle Day 2 or Day 3, a single intra-abdominal injection of Org 36286 180 μg was administered to participants. On stimulation Day 8, a daily subcutaneous dose of Puregon® 150 IU was administered up to and including the time of Pregnyl® administration as a single dose of 10,000 IU subcutaneously. The maximum treatment duration of Puregon® 150 IU was 19 days. Orgalutran® 0.25 mg was administered subcutaneously once daily up to and including the day of Pregnyl®, when the leading follicle reached a size of >= 14 mm.
  Interventions: Drug: Org 36286; Drug: Puregon®; Drug: Orgalutran®; Drug: Pregnyl®
- Org 36286 240 μg + Puregon® 150 IU (Experimental): Cycle Day 2 or Day 3, a single intra-abdominal injection of Org 36286 240 μg was administered to participants. On stimulation Day 8, a daily subcutaneous dose of Puregon® 150 IU was administered up to and including the time of Pregnyl® administration as a single dose of 10,000 IU subcutaneously. The maximum treatment duration of Puregon® 150 IU was 19 days. Orgalutran® 0.25 mg was administered subcutaneously once daily up to and including the day of Pregnyl®, when the leading follicle reached a size of >= 14 mm.
  Interventions: Drug: Org 36286; Drug: Puregon®; Drug: Orgalutran®; Drug: Pregnyl®
- Puregon® 150 IU (Active Comparator): On stimulation Day 8, a daily subcutaneous dose of Puregon® 150 IU was administered up to and including the time of Pregnyl® administration as a single dose of 10,000 IU subcutaneously. The maximum treatment duration of Puregon® 150 IU was 19 days. Orgalutran® 0.25 mg was administered subcutaneously once daily up to and including the day of Pregnyl®, when the leading follicle reached a size of >= 14 mm.
  Interventions: Drug: Puregon®; Drug: Orgalutran®; Drug: Pregnyl®

INTERVENTIONS:
Drug: Org 36286 — Intra-abdominal injection of Org 36286
  Other Names: Corifollitropin alpha
  Arms: Org 36286 120 μg + Puregon® 150 IU; Org 36286 180 μg + Puregon® 150 IU; Org 36286 240 μg + Puregon® 150 IU
Drug: Puregon® — Subcutaneous Puregon® 150 IU
  Other Names: recFSH
Drug: Orgalutran® — Subcutaneous Orgalutran® 0.25 mg
  Other Names: ganirelix (Ganirelix Acetate Injection)
Drug: Pregnyl® — Subcutaneous Pregnyl® 10,000 IU
  Other Names: human chorionic gonadatropin; hCG

SUMMARY:
The primary objective of this trial was to investigate the appropriate dose of a single injection of Org 36286 to initiate multifollicular growth for the first seven days in a controlled ovarian hyperstimulation (COH) protocol for IVF and IVF/ICSI. After seven days, participants were converted to treatment with Puregon® 150 IU and administration of the GnRH antagonist Orgalutran® to finalize the stimulation cycle. Secondary objectives were the safety (including the absence of antibody formation) and the direct effects of Org 36286 on reproductive functions (steroidogenesis, oocyte maturation, embryo quality and implantation).

DETAILED DESCRIPTION:
This trial was made up of two stages with different designs and was conducted at two clinical trial sites. Stage I was open-label and uncontrolled in a small cohort of women (n=6) to obtain first experience in employing Org 36286 in women meeting all inclusion and none of the exclusion criteria. Based on the results of a previous study, the most appropriate dose was anticipated to be 120 μg Org 36286, which was administered on Cycle Day 2 or 3. After seven days, treatment was continued with a fixed dose of 150 IU Puregon® SC. If the size of the leading follicle was >=14 mm, 0.25 mg Orgalutran® SC once daily was administered concurrently with 150 IU Puregon® up to and including the day of hCG. The maximum total treatment duration was 19 days. Treatment of the first two participants with Org 36286 120 μg, that was expected to be adequate for COH, was cancelled due to disrupted follicular growth beyond Day 7. Therefore, the dose of Org 36286 was adapted from 120 μg to 180 µg. Treatment of the first participants gave an indication of the validity of the anticipated doses to be used in Stage II, the actual dose-finding trial. Stage II was open-label, prospective and randomized, comparing three experimental regimens differing in dose of Org 36286 (120 μg, 180 μg, or 240 μg) with a reference treatment. Post-treatment assessments were completed at the visit two weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for COH and IVF or IVF/ICSI;
* Body mass index (BMI) >=18 and <=29 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Ejaculatory sperm;

Exclusion Criteria:

* History of/or current endocrine abnormality such as polycystic ovary syndrome (PCOS), or polycystic ovaries according to ultrasound scan (USS), (treated) hyperprolactinemia or evidence of ovarian dysfunction;
* More than three unsuccessful COH cycles for IVF since the last established ongoing pregnancy (if applicable);
* History of non- or low ovarian response to FSH/human menopausal gonadotropin (hMG) treatment;
* Any clinically relevant hormone value outside the reference range during the early follicular phase (menstrual Cycle Day 2-7) as measured by the local laboratory (FSH, luteinizing hormone [LH], estradiol [E2], progesterone [P], total testosterone [T], thyroid stimulating hormone [TSH], and prolactin);
* Any clinically relevant abnormal laboratory value;
* Any ovarian and/or abdominal abnormality interfering with ultrasound examination;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts);
* Epilepsy, diabetes, cardiovascular, gastro-intestinal, hepatic, renal, pulmonary, or abdominal disease;
* History or presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Hypersensitivity to Orgalutran® or any of its components;
* Administration of investigational drugs within three months prior to screening.
* Use of hormonal preparations within one month prior to the start of Org 36286 with the exception of thyroid medication.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2001-07-01 (Actual); Primary Completion 2002-10-15 (Actual); Study Completion 2002-10-15 (Actual)

PRIMARY OUTCOMES:
Median Puregon® Dose (IU) Required To Reach Criteria for Administration of Human Chorionic Gonadotropin (hCG) For Induction of Final Oocyte Maturation | Day 8 Up to End of Menstrual Cycle

SECONDARY OUTCOMES:
Number of Participants Experiencing Cancellation of Menstrual Cycle | Up to End of Menstrual Cycle
Number of Cumulus-Oocyte-Complexes Experienced By Participants During One Menstrual Cycle | Up to End of Menstrual Cycle
Number of Good Quality Embryos Obtained | Up to One Menstrual Cycle
Number of Participants With Ongoing Pregnancies | Up to 10 Weeks Following hCG Administration
Number of Participants With Anti-Org 36286 Antibodies | Up to 2 Weeks Following Embryo Transfer
Number of Participants With Abnormal Laboratory Findings | Up to 2 Weeks Following Embryo Transfer
Number of Participants With Abnormal Vital Signs | Up to 2 Weeks Following Embryo Transfer
Number of Participants With Serious Adverse Events (SAEs) | Up to 2 Weeks Following Embryo Transfer

REFERENCES:
- [Result] Devroey P, Fauser BC, Platteau P, Beckers NG, Dhont M, Mannaerts BM. Induction of multiple follicular development by a single dose of long-acting recombinant follicle-Stimulating hormone (FSH-CTP, corifollitropin alfa) for controlled ovarian stimulation before in vitro fertilization. J Clin Endocrinol Metab. 2004 May;89(5):2062-70. doi: 10.1210/jc.2003-031766. PMID 15126522